CLINICAL TRIAL: NCT06264505
Title: Probing Participation in Soft Tissue Sarcoma Research: An Observational Study of Soft Tissue Sarcoma Clinical Trials
Brief Title: Investigative Analysis of Soft Tissue Sarcoma Clinical Trials: An Observational Study
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 55955210
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Soft Tissue Sarcoma
Keywords: soft tissue sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Generally, specific demographic cohorts exhibit higher participation rates in medical research, yet there exists a scarcity of research elucidating the trial attributes impacting the engagement of these particular demographics.

The primary objective of this study is to gather extensive data on the clinical trial experiences of individuals diagnosed with soft tissue sarcoma, with the aim of identifying factors hindering patient enrollment or trial completion.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with soft tissue sarcoma
* Aged ≥ 18 years old and ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Subjects willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examination.

Exclusion Criteria:

* Refusal of consent
* Women of childbearing potential without a negative pregnancy test; or women who are lactating.
* Any serious and/or unstable pre-existing medical disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Soft tissue sarcoma patients who are actively deliberating on joining a clinical trial for their condition but have yet to complete the enrollment and randomization stages.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Rate of patients in soft tissue sarcoma clinical research | 3 months
Number of soft tissue sarcoma study participants who maintain involvement until study finish | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] O'Sullivan B, Davis AM, Turcotte R, Bell R, Catton C, Chabot P, Wunder J, Kandel R, Goddard K, Sadura A, Pater J, Zee B. Preoperative versus postoperative radiotherapy in soft-tissue sarcoma of the limbs: a randomised trial. Lancet. 2002 Jun 29;359(9325):2235-41. doi: 10.1016/S0140-6736(02)09292-9. PMID 12103287
- [Background] Pervaiz N, Colterjohn N, Farrokhyar F, Tozer R, Figueredo A, Ghert M. A systematic meta-analysis of randomized controlled trials of adjuvant chemotherapy for localized resectable soft-tissue sarcoma. Cancer. 2008 Aug 1;113(3):573-81. doi: 10.1002/cncr.23592. PMID 18521899
- [Background] Brugemann D, Lehner B, Kieser M, Krisam J, Hommertgen A, Jaekel C, Harrabi SB, Herfarth K, Mechtesheimer G, Sedlaczek O, Egerer G, Geisbusch A, Uhl M, Debus J, Seidensaal K. Neoadjuvant irradiation of extremity soft tissue sarcoma with ions (Extrem-ion): study protocol for a randomized phase II pilot trial. BMC Cancer. 2022 May 12;22(1):538. doi: 10.1186/s12885-022-09560-x. PMID 35550036

DOCUMENTS (1):
  • Informed Consent Form (2024-02-09): https://cdn.clinicaltrials.gov/large-docs/05/NCT06264505/ICF_000.pdf